CLINICAL TRIAL: NCT05274399
Title: The Correlation Between The Hopelessness Level and Self-Care Agency In Patients Receiving Hemodialysis Treatment
Brief Title: Hopelessness and Self-care Power in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Cihat Demirel, Lecturer, Muş Alparslan University
Other Study IDs: E.1337
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Hemodialysis; Despondency; Relational Problems
Keywords: hemodialysis; hopelessness; self-care agency; nurse
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodialysis Patients: Receiving hemodialysis treatment for at least three months
  Interventions: Other: surveys and questionnaires

INTERVENTIONS:
Other: surveys and questionnaires — The data containing the questions determining the relationship between the self-care power and hopelessness of the patients who voluntarily participated in the study were collected through a questionnaire.

SUMMARY:
The purpose of this study is to investigate the correlation between hopelessness level and self-care agency in patient receiving hemodialysis treatment.

DETAILED DESCRIPTION:
While the symptoms and signs that occur as a result of renal failure can be controlled with hemodialysis treatment, the reasons such as the nature of the disease, disease-related symptoms, treatment period and patients' dependency on the hemodialysis machine due to this treatment lead to many physical and psychological problems in the patients. Patients undergoing hemodialysis face physical problems such as becoming dependent, impairment of the socio-economic status, inability to fulfill their role in the society, and changes in work life and various psychological problems such as anxiety, depression, isolation, rejection of the disease, delusions, and hallucinations. it is hoped that this study aiming to determine whether or not there is a correlation between hopelessness level and self-care agency of hemodialysis patients would make a great contribution to the limited available literature.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* To be receiving hemodialysis treatment for at least three months,
* Not having mental confusion or having any psychiatric problems,
* Hearing-sight (except for those who use glasses)-speech problem
* Volunteering to participate in the research

Exclusion Criteria:

* Being 18 years or younger,
* have cognitive impairments,
* not being able to complete the questionnaires,
* not wanting to participate in the study,
* having decided to leave the job

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of 75 patients registered in the hemodialysis unit of this university hospital, and the sample of the study consisted of 69 patients who were treated in this hospital and voluntarily accepted to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | one week after obtaining permission from the institution
  Age, gender, marital status, educational status, employment status, occupation, income level, family type, disease characteristics; Duration of hemodialysis treatment, presence of other chronic diseases, family history of kidney disease, weekly hemodialysis duration (daytime)
Beck Hopelessness Scale (BHS) | one week after obtaining permission from the institution
  Beck Hopelessness Scale (BUS), to determine the level of pessimism about the future of the individual for the purpose of It consists of 20 items expressed as yes and no.
Self-Care Agency Scale | one week after obtaining permission from the institution
  It consists of 22 items scored between 0-2 in order to evaluate the self-care status of patients receiving long-term dialysis treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: no time limit
Access Criteria: All data

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT05274399/SAP_000.pdf